CLINICAL TRIAL: NCT01257932
Title: Monitoring and Predicting Breast Cancer Neoadjuvant Chemotherapy Response Using Diffuse Optical Spectroscopic Imaging
Status: Withdrawn | Type: Observational
Why Stopped: According to the NIH definition of clinical trial studies, this study does not meet requirement to be a clinical trial study.
Sponsor: University of California, Irvine (Other)
Collaborators: American College of Radiology Imaging Network (Network); Massachusetts General Hospital (Other); University of Pennsylvania (Other); Dartmouth-Hitchcock Medical Center (Other); University of San Francisco (Other); M.D. Anderson Cancer Center (Other); Boston University (Other); Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Bruce Tromberg, PhD., Director, Beckman Laser Institute and Medical Clinic, Professor, Departments of Biomedical Engineering and Surgery, University of California, Irvine
Other Study IDs: 20107812
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diagnostic Tool: Diffuse Optical Spectroscopy Imaging Breast Cancer Response to Neoadjuvant Chemotherapy
  Interventions: Device: Diffuse Optical Spectroscopy Imaging

INTERVENTIONS:
Device: Diffuse Optical Spectroscopy Imaging — Diffuse Optical Spectroscopy Imaging Breast Cancer Response to Neoadjuvant Chemotherapy

SUMMARY:
The investigators have developed imaging protocols to monitor and predict breast cancer response to neoadjuvant chemotherapy, both prior to and as early as possible during the course of treatment.

The efficacy and practicality of conventional imaging approaches in the neoadjuvant chemotherapy setting varies and identifies the need for alternate functional imaging strategies. Diffuse optical spectroscopic imaging is an experimental imaging method that allows patients to be followed from baseline through treatment and surgery with a cost-effective, bedside, handheld scanning probe. The researcher evaluates a harmonized diffuse optical spectroscopic imaging technology platform that has been standardized for neoadjuvant chemotherapy monitoring. Diffuse optical spectroscopic imaging is an academic research platform that is non-invasive. Studies will be performed in five clinical sites on approximately 60 neoadjuvant chemotherapy patients.

DETAILED DESCRIPTION:
The investigators are testing the effectiveness of an experimental imaging technology known as Diffuse Optical Spectroscopy Imaging in predicting the success of chemotherapy treatment (shrinkage of tumor).

Diffuse optical spectroscopic imaging measurements are made with a laser breast scanner. This bedside-capable system combines frequency-domain photon migration with steady-state tissue spectroscopy to measure complete(broadband) near-infrared absorption and reduced scattering spectra of breast tissue in vivo. Diffuse Optical Spectroscopy Imaging measurements are made by placing the hand-held probe on the tissue surface and moving the probe to discrete locations along a grid pattern at 1.0 cm intervals. The portable high-bandwidth Frequency-Domain Photon Migration instrument employs intensity-modulated diode lasers and conventional steady-state lamps as sources and an avalanche photodiode as the detector. The time required to perform an Frequency-Domain Photon Migration measurement depends on the desired precision and number of sweeps.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 years of age or older, non pregnant or nursing.
* Diagnosis of breast cancer and will be receiving chemo therapy treatments

Exclusion Criteria:

* 18 years of age or younger, pregnant or nursing.
* Previous treatment including chemo therapy, radiation, surgery, and hormone therapy.
* Previous diagnosis with other form of cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic and community sample
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic Tool Breast Cancer Response to Neoadjuvant Chemotherapy | up to 12 months
  Diffuse Optical Spectroscopy Imaging Breast Cancer Response to Neoadjuvant Chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Tromberg, PhD, Study Director — Beckman Laser Institute
Locations (1):
- Beckman Laser Institute, Irvine, California, United States